CLINICAL TRIAL: NCT01920152
Title: A Randomized Clinical Trial Evaluating Platelet Rich Plasma Versus Hyaluronic-Acid in the Short-term Treatment of Symptomatic OA (Osteoarthritis) of the Hip
Brief Title: Platelet Rich Plasma vs Hyaluronic-Acid in Hip OA (Osteoarthritis)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-0142
Record Dates: First submitted 2013-08-07; First posted 2013-08-09 (Estimated); Results first posted 2021-01-25 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Hip Osteoarthritis
Keywords: Hip, Chondropenia, Osteoarthritis.
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous PRP Hip Injection (Experimental): Patients randomized to this group of treatment will receive 3 blinded hip intra-articular injections of autologous Platelet-Rich Plasma one week apart from each other.
  Interventions: Biological: PRP
- Hyaluronic Acid Hip Injection (Active Comparator): Patients randomized to this group of treatment will receive 3 blinded hip intra-articular injections of hyaluronic acid (SUPARTZ hyaluronate/2.5ml) one week apart each other.
  Interventions: Device: Hyaluronic Acid

INTERVENTIONS:
Biological: PRP — Each PRP preparation requires a total of 36 ml of peripheral blood. This will be obtained via venapuncture and collected in four 9 ml extraction tubes containing 3.8% sodium citrate. The tubes are then centrifuged at 640 rpm for 8 minutes at room temperature. The 1ml plasma fraction located above the buffy coat is aspirated from each tube and dispensed into the fractioning tube. The entire PRP process takes place under laminar airflow. Immediately prior to injection, calcium chloride is is drawn up from the activator ampoule with the activation syringe and is added to the PRP fractioning tube. The activated PRP is then injected in its entirety into the hip joint under strict aseptic technique.
  Arms: Autologous PRP Hip Injection
Device: Hyaluronic Acid — Hyaluronic acid is supplied as a non-pyrogenic solution in 2.5 ml pre-filled syringes and is administered by intra-articular injection using a 22-23 gauge needle. The full 2.5 ml is injected in one joint under strict aseptic administration.
  Other Names: SUPARTZ
  Arms: Hyaluronic Acid Hip Injection

SUMMARY:
The objective of this study is to compare the clinical efficacy of intra-articular injections of autologous platelet rich plasma (PRP) vs hyaluronic acid (HA) for symptomatic early osteoarthritis (OA) of the hip. Secondarily, this study aims to determine the feasibility and safety of treating early OA of the hip with HA and PRP.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a common, painful condition affect adults and causes mobility disability in the United States and Europe. Unfortunately, there is no agents available that halt OA progression. Analgesics and nonsteroidal anti-inflammatory drugs (NSAIDs) have suboptimal effectiveness, and there is concern of systemic side effects.

A large challenge is the development of appropriate and effective therapy in patients with OA. Currently, the most suitable route for administering OA therapy appears to be intra-articular injections that allow accumulation of critical doses of the drug within the damaged area and also reduce the risk of systemic side effects.

The primary objective of this study is to compare the clinical efficacy of intra-articular injections of Platelet Rich Plasma (PRP) vs. Hyaluronic Acid for symptomatic early OA of the hip. Secondarily, the study aims to evaluate the safety and feasibility of both medications delivered.

Patients, which meet inclusion criteria, are confirmed eligible, and agree to enroll in the study, would be randomized and treated with either three intra-articular PRP injections or three intra-articular Hyaluronic Acid injections. If the patient has OA in both hips, they will be randomized to receive the same injection in both hips. The Primary investigator will be unblinded to the treatment that the subject is randomized to. The PI will only be involved in the initial assessment of the patient and the actual injections. All of the follow up visits, clinical assessments and outcome scores will be performed by the sub-investigator, who will also be the examining physician. The sub-investigator will be blinded to the treatment throughout the study. All of the study subjects will be blinded to which treatment that they are assigned to.

Physical exams will be performed to assess range of motion of the hip joint. The difference in ranges of motion will be statistically compared at different time points between the two groups to determine the difference in improvement between the two compared to baseline.

The primary efficacy outcome will be defined as the percentage of patients having a 50% decrease in the summed score for the WOMAC pain subscale from baseline to week 24. We will measure this outcome by applying the WOMAC questionnaire compared with baseline therapy. The secondary efficacy outcomes will also include IHOT and Non Arthritic Hip Score.

An anterior posterior hip radiograph will be performed at 12 months and 24 months to assess Kellgren-Classification and compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 30-72 inclusive.
* Symptomatic early OA of the hip (Kellgren-Lawrence Grade 1-2-3) documented by x-ray taken within the past 6 months.
* Women of childbearing potential will be allowed to enroll but must be willing to practice one highly effective method of contraception (oral, injectable or implanted hormonal methods of contraception, placement of an intrauterine device (IUD) or intrauterine system (IUS) condom or occlusive cap with spermicidal foam/gel/film/cream/suppository, male sterilization, or true abstinence) throughout the study.

Exclusion Criteria:

* Patients with polyarticular disease.
* Patients with major conditions such as poorly control diabetes, Cardiac Heart Failure (CHF), Chronic Obstructive Pulmonary Disease (COPD) or untreated depression
* Patients with known blood disorders (Blood disorders (thrombopathy, thrombocytopenia, anemia with hemoglobin <9g/dL).
* Patients who had intra-articular treatment with steroids within 6 months of randomization in this study or received more than 3 previous intra-articular steroid injections to the effected hip.
* Patients who are pregnant or nursing at the time of consent.
* Patients with inflammatory arthritic conditions (e.g. rheumatoid arthritis)
* Non-English speaking patients. (Scores used for evaluation have not been validated in Spanish)
* Patients who had previous hip surgery
* Additional disabilities in any of the lower limbs that would interfere with any of the clinical assessments.
* Chronic use of NSAID (defined as taking NSAID regularly every week for the last 6 months), steroids or chemotherapy drugs
* Treatment with NSAIDs within 2 days prior to randomization in this study
* Patients with a BMI over 30. Due to the fact that this study utilize an injection technique which may be inaccurate in obese subjects.

Ages: 30 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-08; Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omer Mei-Dan, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Hip Preservation Center, Orthopedic Department, Boulder, Colorado, United States

REFERENCES:
- [Background] Mei-Dan O, McConkey MO, Petersen B, McCarty E, Moreira B, Young DA. The anterior approach for a non-image-guided intra-articular hip injection. Arthroscopy. 2013 Jun;29(6):1025-33. doi: 10.1016/j.arthro.2013.02.014. Epub 2013 Apr 13. PMID 23591381
- [Background] Mei-Dan O, Carmont M, Laver L, Mann G, Maffulli N, Nyska M. Intra-articular injections of hyaluronic acid in osteoarthritis of the subtalar joint: a pilot study. J Foot Ankle Surg. 2013 Mar-Apr;52(2):172-6. doi: 10.1053/j.jfas.2012.12.008. Epub 2013 Jan 17. PMID 23333279
- [Background] Mei-Dan O, Carmont MR, Laver L, Mann G, Maffulli N, Nyska M. Platelet-rich plasma or hyaluronate in the management of osteochondral lesions of the talus. Am J Sports Med. 2012 Mar;40(3):534-41. doi: 10.1177/0363546511431238. Epub 2012 Jan 17. PMID 22253252
- [Background] Mei-Dan O, Laver L, Nyska M, Mann G. [Platelet rich plasma--a new biotechnology for treatment of sports injuries]. Harefuah. 2011 May;150(5):453-7, 490. Hebrew. PMID 21678642
- [Background] Mei-Dan O, Lippi G, Sanchez M, Andia I, Maffulli N. Autologous platelet-rich plasma: a revolution in soft tissue sports injury management? Phys Sportsmed. 2010 Dec;38(4):127-35. doi: 10.3810/psm.2010.12.1835. PMID 21150152
- [Derived] Kraeutler MJ, Houck DA, Garabekyan T, Miller SL, Dragoo JL, Mei-Dan O. Comparing Intra-articular Injections of Leukocyte-Poor Platelet-Rich Plasma Versus Low-Molecular Weight Hyaluronic Acid for the Treatment of Symptomatic Osteoarthritis of the Hip: A Double-Blind, Randomized Pilot Study. Orthop J Sports Med. 2021 Jan 20;9(1):2325967120969210. doi: 10.1177/2325967120969210. eCollection 2021 Jan. PMID 33786329

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from current patient population or first-time patients of the Hip Preservation Clinic or the Joint Clinic between 2013 and 2018. Participants were identified and recruited during routine office visits. The first participant was enrolled on December 5th, 2013 and the last participant was enrolled in December 2017.
Pre-assignment Details: There were 63 participants assessed for eligibility. Of the 38 enrolled participants, 34 participants (36 hips) met the inclusion criteria and were randomized to treatment.
Units Other Than Participants: Hips
Groups:
- Autologous PRP Hip Injection: Participants were randomized to this group of treatment. Participants who received 3 blinded hip intra-articular injections of autologous Platelet-Rich Plasma one week apart from each other and completed a minimum 6-week follow-up were included in the study.
  PRP: Each PRP preparation requires a total of 36 ml of peripheral blood. This will be obtained via venapuncture and collected in four 9 ml extraction tubes containing 3.8% sodium citrate. The tubes are then centrifuged at 640 rpm for 8 minutes at room temperature. The 1ml plasma fraction located above the buffy coat is aspirated from each tube and dispensed into the fractioning tube. The entire PRP process takes place under laminar airflow. Immediately prior to injection, calcium chloride is is drawn up from the activator ampoule with the activation syringe and is added to the PRP fractioning tube. The activated PRP is then injected in its entirety into the hip joint under strict aseptic technique.
- Hyaluronic Acid Hip Injection: Participants were randomized to this group of treatment. Participants who received 3 blinded hip intra-articular injections of hyaluronic acid (SUPARTZ hyaluronate/2.5ml) one week apart each other and completed a minimum 6-week follow-up were included in the study.
  Hyaluronic Acid: Hyaluronic acid is supplied as a non-pyrogenic solution in 2.5 ml pre-filled syringes and is administered by intra-articular injection using a 22-23 gauge needle. The full 2.5 ml is injected in one joint under strict aseptic administration.
Period: Overall Study
Arm/Group | Autologous PRP Hip Injection | Hyaluronic Acid Hip Injection
Started | 19; 20 Hips | 15; 16 Hips
Completed | 18; 19 Hips | 13; 14 Hips
Not Completed | 1; 1 Hips | 2; 2 Hips
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: The Hyaluronic Acid Hip Injection group comprised 13 patients (14 hips) and the Autologous PRP Hip Injection group comprised 18 patients (19 hips). Two patients underwent bilateral treatments, one in each group.
Units Other Than Participants: Hips
Groups:
- Total: Total of all reporting groups
Arm/Group | Autologous PRP Hip Injection | Hyaluronic Acid Hip Injection | Total
Number analyzed (Participants) | 18 | 13 | 31
Number analyzed (Hips) | 19 | 14 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] — The Hyaluronic Acid Hip Injection group comprised 13 patients (14 hips) and the Autologous PRP Hip Injection group comprised 18 patients (19 hips). Two patients underwent bilateral treatments, one in each group.
  Age (at the time of the first hip injection) is presented for the hips, rather than the patients. Therefore, patients with data for two hips were included, and their age was counted twice.
  years | 53.3 (8.4) | 54.5 (9.0) | 53.8 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 13
  Male | 8 | 10 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 12 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 18 | 13 | 31
BMI [Mean (Standard Deviation); unit: Kg/m^2] — The Hyaluronic Acid Hip Injection group comprised 13 patients (14 hips) and the Autologous PRP Hip Injection group comprised 18 patients (19 hips). Two patients underwent bilateral treatments, one in each group.
  BMI (at the time of the first hip injection) is presented for the hips, rather than the patients. Therefore, patients with data for two hips were included, and their BMI was counted twice.
  Kg/m^2 | 23.7 (2.1) | 23.5 (2.0) | 23.6 (2.0)
Kellgren-Lawrence (KL) Grading Scale [Count of Units; unit: Hips] — Anterior posterior hip x-rays were performed at baseline for each hip and classified according to Kellgren-Lawrence (KL) grading scale: 0 = normal; 1 = doubtful narrowing of joint space and possible osteophytic lipping; 2 = definite osteophytes and possible narrowing of joint space; 3 = moderate multiple osteophytes, definite narrowing of joint space, some sclerosis, and possible deformity of bone contour; 4 = large osteophytes, marked narrowing of joint space, severe sclerosis, and definite deformity of bone contour. Possible scores range from 0-4. Higher scores indicate a worse outcome.
  Hips
    KL Grade 2 | 7 | 2 | 9
    KL Grade 3 | 12 | 12 | 24
    KL Grade 4 | 0 | 0 | 0
    KL Grade 0 | 0 | 0 | 0
    KL Grade 1 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Survivorship, as Measured by the Frequency of Patient Withdrawal of Their Treated Hip to Undergo Surgery (Total Hip Arthroplasty [THA] or Hip Resurfacing Procedure).
Description: To measure duration of clinical benefit, survivorship was analyzed by investigating the frequency of patient withdrawal of their treated hip to undergo surgery (total hip arthroplasty [THA] or hip resurfacing procedure). Survivorship was evaluating hips, not patients in this outcome measure. This served as the primary outcome measure for the study.
Time Frame: Baseline, 24 Months
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Autologous PRP Hip Injection | Hyaluronic Acid Hip Injection
Number analyzed (Participants) | 18 | 13
Number analyzed (Hips) | 19 | 14
Hips | 3 | 7

2. Primary Outcome: Change in Western Ontario and McMaster Universities Arthritis Index (WOMAC) Pain Sub-score
Description: The primary efficacy outcome was defined as the percentage of patients having a 50% decrease in the summed score for the Western Ontario and McMaster Universities Arthritis Index (WOMAC) pain sub-score from baseline to week 24.
  The WOMAC score is a normalized patient-reported outcome measure in which 0 represents the worst possible score and 100 represents the best possible score. The WOMAC is primarily used in osteoarthritis clinical trials to evaluate the effects of arthroplasty and drug interventions in patients with hip osteoarthritis.
  Thus, a 50% increase in the WOMAC pain sub-score would indicate reduced pain or improvement, while a 50% decrease would indicate worsening pain.
Time Frame: Baseline, Week 24
Population: The overall number analyzed decreased in the PRP group due to a participant withdrawing from the study to undergo a total hip replacement at week 12.
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Autologous PRP Hip Injection | Hyaluronic Acid Hip Injection
Number analyzed (Participants) | 17 | 13
Number analyzed (Hips) | 18 | 14
Hips
  ≥50% Decrease in WOMAC Pain (Worse) | 0 | 0
  ≥50% Increase in WOMAC Pain (Better) | 2 | 0

3. Secondary Outcome: Western Ontario and McMaster Universities Arthritis Index (WOMAC) Scores at Baseline
Description: The Western Ontario and McMaster Universities Arthritis Index (WOMAC) score was defined as the secondary outcome measurement. The WOMAC score is a normalized patient-reported outcome measure in which 0 represents the worst possible score and 100 represents the best possible score. The WOMAC is primarily used in osteoarthritis clinical trials to evaluate the effects of arthroplasty and drug interventions in patients with hip osteoarthritis.
Time Frame: Baseline
Population: The number analyzed for some of the WOMAC subscores differs from the overall number analyzed due to item non-response.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Hips
Arm/Group | Autologous PRP Hip Injection | Hyaluronic Acid Hip Injection
Number analyzed (Participants) | 18 | 13
Number analyzed (Hips) | 19 | 14
score on a scale
  WOMAC Pain | 72.1 (18.0) | 78.9 (14.3)
  WOMAC Joint | 55.3 (26.5) | 68.8 (24.9)
  WOMAC Function: number analyzed (Participants) | 17 | 12
  WOMAC Function: number analyzed (Hips) | 18 | 13
  WOMAC Function | 69.6 (20.4) | 81.2 (12.9)
  WOMAC Overall: number analyzed (Participants) | 17 | 12
  WOMAC Overall: number analyzed (Hips) | 18 | 13
  WOMAC Overall | 67.6 (19.7) | 77.9 (14.4)

4. Secondary Outcome: Western Ontario and McMaster Universities Arthritis Index (WOMAC) Scores at Week 6
Description: as for outcome 3
Time Frame: Week 6
Population: The number analyzed for some of the WOMAC subscores differs from the overall number analyzed due to item non-response.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Hips
Arm/Group | Autologous PRP Hip Injection | Hyaluronic Acid Hip Injection
Number analyzed (Participants) | 18 | 13
Number analyzed (Hips) | 19 | 14
score on a scale
  WOMAC Pain: number analyzed (Participants) | 17 | 11
  WOMAC Pain: number analyzed (Hips) | 18 | 12
  WOMAC Pain | 80.8 (12.4) | 80.0 (17.1)
  WOMAC Joint: number analyzed (Participants) | 17 | 12
  WOMAC Joint: number analyzed (Hips) | 18 | 13
  WOMAC Joint | 71.5 (15.9) | 75.0 (23.4)
  WOMAC Function: number analyzed (Participants) | 17 | 13
  WOMAC Function: number analyzed (Hips) | 18 | 14
  WOMAC Function | 82.9 (12.5) | 83.7 (15.2)
  WOMAC Overall: number analyzed (Participants) | 17 | 11
  WOMAC Overall: number analyzed (Hips) | 18 | 12
  WOMAC Overall | 79.7 (10.9) | 79.5 (16.2)

5. Secondary Outcome: Western Ontario and McMaster Universities Arthritis Index (WOMAC) Scores at Week 12
Description: as for outcome 3
Time Frame: Week 12
Population: The number analyzed for some of the WOMAC subscores differs from the overall number analyzed due to item non-response of a participant who underwent bilateral treatment in the HA group. The overall number analyzed decreased in the PRP group due to a participant withdrawing from the study to undergo a total hip replacement at week 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Hips
Arm/Group | Autologous PRP Hip Injection | Hyaluronic Acid Hip Injection
Number analyzed (Participants) | 17 | 13
Number analyzed (Hips) | 18 | 14
score on a scale
  WOMAC Pain: number analyzed (Hips) | 18 | 13
  WOMAC Pain | 80.8 (12.0) | 79.2 (18.0)
  WOMAC Joint: number analyzed (Hips) | 18 | 13
  WOMAC Joint | 68.8 (19.8) | 71.2 (29.2)
  WOMAC Function: number analyzed (Hips) | 18 | 13
  WOMAC Function | 80.1 (14.8) | 79.1 (17.8)
  WOMAC Overall: number analyzed (Hips) | 18 | 13
  WOMAC Overall | 78.0 (13.0) | 77.5 (19.0)

6. Secondary Outcome: Western Ontario and McMaster Universities Arthritis Index (WOMAC) Scores at Week 24
Description: as for outcome 3
Time Frame: Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Hips
Arm/Group | Autologous PRP Hip Injection | Hyaluronic Acid Hip Injection
Number analyzed (Participants) | 17 | 13
Number analyzed (Hips) | 18 | 14
score on a scale
  WOMAC Pain | 76.1 (15.1) | 84.3 (14.5)
  WOMAC Joint | 72.9 (22.8) | 74.1 (22.2)
  WOMAC Function | 80.2 (16.4) | 84.1 (15.7)
  WOMAC Overall | 77.0 (15.8) | 82.1 (15.1)

7. Secondary Outcome: Change in Western Ontario and McMaster Universities Arthritis Index (WOMAC) Scores
Description: as for outcome 3
Time Frame: Baseline, Month 24
Population: Fourteen participants (15 hips, 74%) in the PRP group reached a final follow-up of 24 months. Five participants (5 hips, 36%) in the HA group reached a final follow-up of 24 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Hips
Arm/Group | Autologous PRP Hip Injection | Hyaluronic Acid Hip Injection
Number analyzed (Participants) | 14 | 5
Number analyzed (Hips) | 15 | 5
score on a scale
  WOMAC Pain | 6.67 (15.99) | 0 (18.37)
  WOMAC Joint | 12.5 (28.74) | -2.5 (16.3)
  WOMAC Function | 9.81 (16.45) | -2.65 (18.67)
  WOMAC Overall | 9.05 (17.88) | -1.51 (14.14)

8. Secondary Outcome: Hip Range of Motion (ROM) at Baseline
Description: The range of motion (ROM) of the hip is reported for both groups of treatment. This includes external rotation (ER), internal rotation (IR), and flexion (FL).
Time Frame: Baseline
Population: The number analyzed differs from the overall number analyzed due to missing data. It is important to note that some patients were unable to reach 0 degrees of hip IR and therefore the value was recorded as negative.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Hips
Arm/Group | Autologous PRP Hip Injection | Hyaluronic Acid Hip Injection
Number analyzed (Participants) | 18 | 13
Number analyzed (Hips) | 19 | 14
degrees
  IR: number analyzed (Participants) | 17 | 13
  IR: number analyzed (Hips) | 18 | 14
  IR | 2.8 (7.0) | 2.3 (13.5)
  ER: number analyzed (Participants) | 17 | 13
  ER: number analyzed (Hips) | 18 | 14
  ER | 36.1 (12.9) | 36.4 (10.8)
  FL: number analyzed (Participants) | 17 | 13
  FL: number analyzed (Hips) | 18 | 14
  FL | 102.4 (8.2) | 101.1 (11.3)

9. Secondary Outcome: Hip Range of Motion (ROM) at Week 6
Description: as for outcome 8
Time Frame: Week 6
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Hips
Arm/Group | Autologous PRP Hip Injection | Hyaluronic Acid Hip Injection
Number analyzed (Participants) | 18 | 13
Number analyzed (Hips) | 19 | 14
degrees
  IR: number analyzed (Participants) | 17 | 12
  IR: number analyzed (Hips) | 18 | 13
  IR | 3.3 (6.6) | 0.9 (14.1)
  ER: number analyzed (Participants) | 17 | 12
  ER: number analyzed (Hips) | 18 | 13
  ER | 37.6 (9.2) | 36.2 (9.2)
  FL: number analyzed (Participants) | 17 | 12
  FL: number analyzed (Hips) | 18 | 13
  FL | 99.6 (7.8) | 99.2 (9.8)

10. Secondary Outcome: Hip Range of Motion (ROM) at Week 12
Description: as for outcome 8
Time Frame: Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Hips
Arm/Group | Autologous PRP Hip Injection | Hyaluronic Acid Hip Injection
Number analyzed (Participants) | 18 | 13
Number analyzed (Hips) | 19 | 14
degrees
  IR: number analyzed (Participants) | 17 | 13
  IR: number analyzed (Hips) | 18 | 14
  IR | 4.7 (7.9) | 0.7 (14.5)
  ER: number analyzed (Participants) | 17 | 13
  ER: number analyzed (Hips) | 18 | 14
  ER | 34.6 (12.2) | 35.7 (8.7)
  FL: number analyzed (Participants) | 17 | 13
  FL: number analyzed (Hips) | 18 | 14
  FL | 101.9 (12.2) | 98.2 (9.3)

11. Secondary Outcome: Hip Range of Motion (ROM) at Week 24
Description: as for outcome 8
Time Frame: Week 24
Population: The number analyzed differs from the overall number analyzed due to missing data. The overall number analyzed decreased in the PRP group due to a participant withdrawing from the study to undergo a total hip replacement at week 12.
  It is important to note that some patients were unable to reach 0 degrees of hip IR and therefore the value was recorded as negative.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Hips
Arm/Group | Autologous PRP Hip Injection | Hyaluronic Acid Hip Injection
Number analyzed (Participants) | 17 | 13
Number analyzed (Hips) | 18 | 14
degrees
  IR: number analyzed (Participants) | 17 | 12
  IR: number analyzed (Hips) | 18 | 13
  IR | 7.8 (10.3) | 0.8 (11.3)
  ER: number analyzed (Participants) | 17 | 12
  ER: number analyzed (Hips) | 18 | 13
  ER | 36.8 (10.1) | 38.5 (7.5)
  FL: number analyzed (Participants) | 17 | 12
  FL: number analyzed (Hips) | 18 | 13
  FL | 103.5 (13.3) | 97.3 (10.1)

12. Secondary Outcome: Change in Hip Range of Motion (ROM)
Description: as for outcome 8
Time Frame: Baseline, 24 Months
Population: Fourteen participants (15 hips, 74%) in the PRP group reached a final follow-up of 24 months. Five participants (5 hips, 36%) in the HA group reached a final follow-up of 24 months.
  It is important to note that some patients were unable to reach 0 degrees of hip IR and therefore the value was recorded as negative.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Hips
Arm/Group | Autologous PRP Hip Injection | Hyaluronic Acid Hip Injection
Number analyzed (Participants) | 14 | 5
Number analyzed (Hips) | 15 | 5
degrees
  IR | 3.36 (7.88) | 2.6 (9.29)
  ER | -0.3571 (13.65) | 0 (11.73)
  FL | -2.5 (8.49) | 0 (5)

13. Secondary Outcome: Change in International Hip Outcome Tool (IHOT)
Description: The International Hip Outcome Tool (IHOT) score is reported for both groups of treatment as the change from baseline to 24 months post-injection.
  The iHOT12 instrument is a joint-specific PRO for evaluating quality of life (QoL). A score of 100 indicates excellent QoL (full function and no symptoms), whereas zero signifies the worst QoL (maximum limitations and extreme symptoms).
Time Frame: Baseline, 24 Months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Hips
Arm/Group | Autologous PRP Hip Injection | Hyaluronic Acid Hip Injection
Number analyzed (Participants) | 14 | 5
Number analyzed (Hips) | 15 | 5
score on a scale | 20.61 (22.59) | -3.92 (18.68)

14. Secondary Outcome: Change in Non-Arthritic Hip Score
Description: The Non Arthritic Hip subjective score is reported for both groups of treatment as the change from baseline to 24 months post-injection.
  The maximum score is 100 indicating normal hip function.
Time Frame: Baseline, 24 Months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Hips
Arm/Group | Autologous PRP Hip Injection | Hyaluronic Acid Hip Injection
Number analyzed (Participants) | 14 | 5
Number analyzed (Hips) | 15 | 5
score on a scale | 6.09 (23.97) | -7.26 (15.97)

15. Secondary Outcome: Change in Flexion-Abduction-External Rotation (FABER) Test.
Description: The flexion-abduction-external rotation (FABER) test is a clinical test utilized as a provocation test to detect hip, lumbar spine, or sacroiliac joint pathology. A positive FABER test is one that reproduces the patient's pain or limits their range of movement, while a negative FABER test is one that does not reproduce the patient's pain or limit their range of movement.
  The FABER test is reported for both groups of treatment as count of hips experiencing a decrease in pain (from a positive test to a negative test) during the FABER test from baseline to 24 months.
Time Frame: Baseline, 24 Months
Population: as for outcome 7
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Autologous PRP Hip Injection | Hyaluronic Acid Hip Injection
Number analyzed (Participants) | 14 | 5
Number analyzed (Hips) | 15 | 5
Hips | 7 | 3

16. Secondary Outcome: Change in Anterior Posterior (AP) Pelvis Radiograph/ Kellgren-Lawrence Grading Scale Classification.
Description: Anterior posterior hip x-rays were performed for each hip and classified according to Kellgren-Lawrence (KL) grading scale, which is defined as follows:
  0 = normal; 1 = doubtful narrowing of joint space and possible osteophytic lipping; 2 = definite osteophytes and possible narrowing of joint space; 3 = moderate multiple osteophytes, definite narrowing of joint space, some sclerosis, and possible deformity of bone contour; 4 = large osteophytes, marked narrowing of joint space, severe sclerosis, and definite deformity of bone contour.
  The Kellgren-Lawrence (KL) Grading Scale is reported for both groups of treatment as the change from baseline to 24 months.
Time Frame: Baseline, 24 Months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Hips
Arm/Group | Autologous PRP Hip Injection | Hyaluronic Acid Hip Injection
Number analyzed (Participants) | 14 | 5
Number analyzed (Hips) | 15 | 5
score on a scale | 0.5 (0.6) | 0.6 (0.5)

17. Other Pre Specified Outcome: Number of Patients With Adverse Events
Description: Type, duration and trend of every adverse event for each patient will be reported
Time Frame: Week 2-Week 3 and 6-12-18-24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The nature, onset, duration, severity, and outcome of all adverse events, as well as any association of an adverse event related to the study medication, was assessed and documented at each visit (Week 1, Week 2, Week 3, Week 6, Month 3, Month 6, Month 12, Month 18, Month 24).
Arm/Group | Autologous PRP Hip Injection | Hyaluronic Acid Hip Injection
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/15
Other Adverse Events (participants affected / at risk) | 0/19 | 0/15

LIMITATIONS AND CAVEATS:
Outcome measures descriptions are accurate to the approved protocol. Wording was modified slightly from the original registration for the purposes of results data reportability to the ClinicalTrials.gov data tables.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT01920152/Prot_SAP_000.pdf